CLINICAL TRIAL: NCT03952195
Title: Ileal Pouch Salvage and Excision Operations: Indications, Complications and Outcomes
Brief Title: Complications and Outcomes of Pouch Excision
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joel Bauer, Professor of Surgery, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 16-0172
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: IPAA; IBD; Ulcerative Colitis; Restorative Proctocolectomy; Ileal Pouch-Anal Anastomosis; Excisions; Salvage; Pouch
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Procedure is offered today to most patients with chronic ulcerative colitis (CUC) or familial adenomatous polyposis (FAP) who are candidates for total proctocolectomy. While high rates of successful pouch surgery are reported, there is a significant long-term risk of pouch-related complications including ileo-anal anastomotic separation and stricture, pouch-perineal and pouch-vaginal fistula, pouchitis, pelvic sepsis, small bowel obstruction, and pouch dysfunction. Despite recent advances in treatment of these complications by medical and surgical means, these problems can still lead to pouch failure and pouch excision. The long-term rate of pouch excision is reported in large series to range from 5.3% to 24%. Moreover, the burden of quality of life impairment on patients with these complications is immense. Pouch excision operations are technically difficult with substantial morbidity. This study aimed to investigate the indications for pouch excision, the number of salvage operations prior to these excisions and complications of pouch excision surgeries.

DETAILED DESCRIPTION:
Data Collection Data were collected by retrospective review of a single institution, single practice, prospectively maintained clinical database consisting of 1263 patients undergoing RPC with IPAA performed between 1981 and 2015. All cases of pouch excision were identified. The recorded data comprised of patient demographic details, pathologic diagnoses at the time of pouch formation and pouch excision, details on the surgical procedures performed including formation of the pouch, procedures performed attempting to salvage the pouch, excision of the pouch, and intraoperative and early (within 30 days after pouch excision surgery) complications.

Pouch Salvage Surgery The type and date of all pouch salvage surgical interventions performed under general anesthesia prior to pouch excision were documented and categorized. We documented and classified each trip to the operating room as a salvage encounter. Salvage procedures were defined as any surgical intervention performed to preserve the pouch and did not include procedures unrelated to the pouch, such as incisional hernia repairs. Operative salvage procedures included abscess drainage with incision and drainage of an abscess cavity and curettage of peri-pouch abscesses or fistula tracts. Fistula repair included any repair of peri-pouch fistulae including seton placement and advancement flap. Any transanal or abdominal repair or revision of the pouch including the pouch-anal anastomosis was classified as a pouch revision. Diversion was defined as the formation of any unplanned diverting loop ileostomy. Ileostomy reversal was defined as the restoration of continuity following an unplanned diversion. Loop ileostomies formed or reversed as part of a planned, staged RPC procedure were excluded. Other procedures included dilatation of the IPAA anastomosis with examination under anesthesia (EUA), formation of an entero-pouch bypass, and any resections of peri-pouch cysts or desmoids.

Indications for Pouch Excision Indications for pouch excision were based on documented preoperative clinical and histopathologic diagnoses. Pouch dysfunction was defined as stool incontinence with or without obstructed defecation. Pouchitis was separately defined as clinical symptoms of bleeding, cramping abdominal pain, anal discharge, tenesmus, urgency, and increased frequency of defecation [10]. Distinguishing between pouchitis and pouch dysfunction was based on the operating surgeon's preoperative clinical diagnosis rather than pathology. Septic complications included any pelvic, perineal, or perianal infection as a result of anastomotic dehiscence, abscess or persistent fistula arising from the pouch or IPAA. Other indications for pouch excision included cancer diagnosed from endoscopic biopsy or found at surgery. Pouch necrosis was defined as complete transmural ischemia of the pouch.

Summary Measures and Statistical Analyses. Summary statistics of continuous variables reported the mean and standard deviation (SD) and the median and interquartile range (IQR) as appropriate. Pouch survival was defined as the time between pouch formation and pouch excision surgeries. The rate of salvage encounters was calculated by the sum of all encounters in the operating room where the primary surgery was to salvage the pouch divided by the number of patients. Differences in pouch survival by indication for pouch excision were compared using log-rank test. Statistical significance was defined as P<0.05.

Excluded and Missing Data Missing data were not included in the analyses. One patient with FAP had her pouch formed in our center, sought care at an outside institution for her pouch excision and the indication for pouch excision was unknown. However, data collected at the time of pouch formation and salvage procedures performed on this patient prior to excision were available and included in the analyses. Another patient developed pouch necrosis two weeks after pouch formation surgery, the pouch was never functional, and this patient was not included in our analyses of pouch survival or salvage encounter rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pouch excision

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had an their pouch excised
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with complications | Five years
  Number of Participants with any post operative complication

CONTACTS AND LOCATIONS:
Overall Officials: Joel J Bauer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No